CLINICAL TRIAL: NCT07025720
Title: Personalized Accelerated TMS for High-Risk Adolescent Depression
Acronym: PATH-RAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Sorensen Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2227384
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder (MDD); Suicidal Ideation
Keywords: TMS; MDD; Suicidal ideation; transcranial magnetic stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TMS (Experimental)
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — The protocol involves delivering sessions of intermittent theta burst stimulation (iTBS) of 60 cycles of 10 bursts of three pulses at 50 Hz were delivered in 2-second trains (5 Hz) with an 8-second intertrain interval. Stimulation sessions will be delivered hourly. Ten sessions will be applied per day (18,000 pulses/day) for 5 consecutive days (90,000 pulses in total). Stimulation will be delivered at 90% resting motor threshold (rMT) adjusted for cortical depth.
  MR brain imaging will be used with the Localite Neuronavigation System (Localite GmbH, Sankt Augustin, Germany) to position the TMS coil over the individualized stimulation target.

SUMMARY:
The goal of this clinical trial is to learn if a fast-acting brain stimulation treatment called transcranial magnetic stimulation (TMS) can help people with depression and suicidal thoughts. The treatment is non-invasive (does not involve surgery or medications), is given over 5 days, and uses brain imaging (MRI) to guide which part of the brain to target. This study tests whether this treatment is a helpful and practical option for adolescents and young adults who are depressed and have suicidal thoughts.

We want to see if:

1. This treatment is feasible and acceptable to patients
2. It can reduce depression and suicidal thoughts
3. It can lower the chance of going to the hospital
4. It affects daily functioning (school, work, relationships)

All participants will undergo 5-days of TMS treatment and complete MRI brain scans before and after treatment. They will return for check-ups after 1 week and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Able to provide informed consent
* age 15 years or older
* Discharged within the past week from the ED for chief complaint of SI OR recently admitted in urgent health care setting or seen in outpatient clinic for depression-related suicidal ideation
* Meets MDD criteria per the Mini International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

* Unable to consent (due to medical condition, psychosis, substance use, etc)
* Use of benzodiazepines or medications that would interfere with TMS treatment as per PI discretion
* Active substance use or severe substance use that in the opinion of the PI would interfere with study participation
* Untreated, active psychosis
* Female patient who is breastfeeding, pregnant or who is planning a pregnancy during the study
* Participation in any clinical study with exposure to any investigational treatment or product within the previous 30 days, or plan on concurrent participation in other studies
* Contraindications to receiving TMS and/or MRI as determined by screening questionnaires

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in MADRS score | 1 week
  Change in depressive symptoms as measured by The Montgomery-Åsberg Depression Rating Scale (MADRS) from baseline to post-rTMS treatment. MADRS scores range from 0 to 60, with higher scores reflecting greater severity of depressive symptoms.

SECONDARY OUTCOMES:
Change in C-SSRS score | 1 week
  Change in suicidal ideations as measured by Columbia Suicide Severity Rating Scale (C-SSRS) from baseline to post-treatment. Suicidal ideation is assessed using a 5-point scale (range: 0-5), with higher scores indicating greater severity.
Health utilization rate | 1 week, 1 month
  Rates of health visits at 1-week and 1 month follow-up
Change in Q_LES_Q_SF score | 1 week and 1 month
  Change in functional impairment as measured by the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q_LES_Q_SF). Scores range from 14 to 70, with higher scores indicating better quality of life

OTHER OUTCOMES:
Changes in Functional Connectivity | 1 week, 1 month
  To explore the changes in functional connectivity patterns associated with the antidepressant and anti-suicidal effects of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided